CLINICAL TRIAL: NCT01080703
Title: Does The Lower Extremity Resistance Program Improve Quadriceps Strength, Endurance, And Quality Life In Pre-Lung Transplant Patients?
Brief Title: To Determine if a Lower Extremity Strengthening Program Improve Quadriceps Muscle Strength
Acronym: Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-076-B; PULMONARY
Record Dates: First submitted 2010-03-02; First posted 2010-03-04 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Pulmonary Disease
Keywords: Lung Transplant; Quadriceps Strength; Quality of Life; Patients with pulmonary disease awaiting lung transplant.
MeSH Terms: conditions — Lung Diseases | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lower extremity strengthening (Experimental)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Lower extremity resistance exercises and aerobic exercises 3 times a week in 10 week pulmonary rehabilitation program prior to lung transplant.

SUMMARY:
The purpose of this study is to determine if a lower extremity strengthening program as part of pulmonary rehabilitation will improve quadriceps muscle strength, endurance and functional status as well as overall quality of life.

Hypothesis:

1. Lower extremity resistance training as part of a pulmonary rehabilitation program will improve quadriceps strength, endurance and functional capacity.
2. Lower extremity resistance training as part of a pulmonary rehabilitation program will improve quality of life in patients awaiting lung transplant.

DETAILED DESCRIPTION:
Objectives:

1. To determine if a lower extremity strengthening program as part of pulmonary rehabilitation is effective at increasing quadriceps strength when measured with a hand held dynamometer.
2. To determine the effectiveness of a lower extremity strengthening program as part of pulmonary rehabilitation for improving endurance and functional capacity as measured by the six minute walk test.
3. To determine if the lower extremity strengthening program as part of pulmonary rehabilitation improves overall quality of life as measured by the St. George's Respiratory Questionnaire.
4. To provide a basic framework for a larger randomized control study evaluating if a lower extremity strengthening program as part of a pulmonary rehabilitation program is more effective than a pulmonary rehabilitation program alone at improving quadriceps strength, endurance, and functional level.

ELIGIBILITY:
Inclusion Criteria:

* Patients preparing for lung transplant
* Diagnoses included are: Chronic Obstructive Pulmonary Disease, Idiopathic Pulmonary Fibrosis, Sarcoidosis, Cystic Fibrosis, or Bronchiectasis

Exclusion Criteria:

* Primary Pulmonary Hypertension
* Multi-organ transplant patients
* Re-transplant patients
* Patients requiring intubation greater than or equal to 7 days prior to transplant
* Any orthopedic condition which will prevent from participation in a lower extremity strengthening program

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Quadriceps Strength | 10 weeks
  Quadriceps Strength will be assessed at initial evaluation and subsequently every two weeks for 10 weeks. Testing will be done at 30, 60 and 90 degrees of knee flexion using hand held dynamometer. The six miute walk test is also used as a primary outcomes to assess endurance. It will be done at initial evaluation, 5 weeks and 10 weeks.

SECONDARY OUTCOMES:
Quality of Life Survey | 10 weeks
  The St. George Respiratory Questionnaire will be used to assess quality of life at initial evaluation and at 10 weeks (completion of program).

CONTACTS AND LOCATIONS:
Overall Officials: Edward R Garrity, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago Medical Center, Chicago, Illinois, United States